CLINICAL TRIAL: NCT01407107
Title: Phase I Dose Escalation Trial of Nitroglycerin in Addition to 5-flourouracil and Radiation Therapy for Neo-adjuvant Treatment of Operable Rectal Cancer
Brief Title: Dose Escalation Trial of Nitroglycerin, 5-flourouracil and Rad Therapy for Rectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jonathan E. Dowell, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 122010-172
Record Dates: First submitted 2011-07-29; First posted 2011-08-01 (Estimated); Results first posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2020-12

CONDITIONS: Rectal Cancer
Keywords: nitroglycerin; 5-flourouracil; radiation therapy; neo-adjuvant treatment
MeSH Terms: conditions — Rectal Neoplasms | interventions — Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nitroglycerin (Experimental): Dose escalation trial of Nitroglycerin
  Interventions: Drug: Nitroglycerin 0.2 MG/HR; Drug: Nitroglycerin 0.4 MG/HR; Drug: Nitroglycerin 0.6 MG/HR

INTERVENTIONS:
Drug: Nitroglycerin 0.2 MG/HR — 0.2mg/hr nitroglycerin transdermal patch daily. The first 3 patients will have a low dose patch applied (0.2 mg/hr).
Drug: Nitroglycerin 0.4 MG/HR — 0.4mg/hr nitroglycerin transdermal patch daily. The first 3 patients will have a low dose patch applied (0.2 mg/hr) if this is well tolerated a higher dose patch (0.4mg/hr) will be used for the next 3 patients.
Drug: Nitroglycerin 0.6 MG/HR — 0.6mg/hr nitroglycerin transdermal patch daily. The first 3 patients will have a low dose patch applied (0.2 mg/hr) if this is well tolerated a higher dose patch (0.4mg/hr) will be used for the next 3 patients and if this is well tolerated an even higher dose patch (0.6mg/hr) will be used.

SUMMARY:
The purpose of this study is to determine whether topical nitroglycerin in addition to 5-flourouracil and radiation therapy are effective in the treatment of operable rectal cancer.

DETAILED DESCRIPTION:
This is an open label, non-randomized, multi-cohort, dose escalation trial to evaluate the safety, tolerability, feasibility and maximum tolerated dose (MTD) of topical nitroglycerin in addition to 5-flourouracil and radiation therapy for neo-adjuvant treatment of, T3-T4 or clinically node positive, operable rectal cancer.

Patients that would otherwise be eligible for concurrent neo-adjuvant chemotherapy with continuous infusion 5-FU, for locally advanced operable rectal cancer, will be assigned to 4 sequential cohorts of 3 different dose levels of nitro glycerin patches (0.2; 0.4; and 0.6 mg/hr). Each cohort will consist of 3 patients. All patients will receive radiation therapy, 45-50 Gy in 25-28 fractions to the pelvis along with continuous infusion 5-FU 225mg/M2 for the duration of the radiation therapy. The radiation therapy will be planned and delivered as per institutional standard of care for the Dallas VAMC radiation oncology department.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven Rectal Adenocarcinoma
* Histological diagnosis of operable T3-4, or T1-4 node positive, M0 rectal adenocarcinoma using endorectal ultrasound and/or MRI in addition to Computed Tomography (CT) of the chest, abdomen and pelvis for pre-study staging Acceptable alternatives for systemic staging instead of CT chest , abdomen, pelvis are CT abdomen and pelvis plus a Chest X-ray or a PET/CT
* Ability to give informed consent and willingness to adhere to study protocol
* Age ≥ 18 years and otherwise eligible to receive medical care at the Dallas VA Medical Center.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Adequate hematological, hepatic and renal function defined as in protocol.

Exclusion Criteria:

* Any condition that would hamper informed consent or ability to comply with the study protocol
* Significant history of cardiac disease, e.g. uncontrolled hypertension, unstable angina, decompensated congestive-heart failure, myocardial infarction within the last six months or ventricular arrhythmias requiring medication.
* Pregnant and lactating women.
* Patients taking Phosphodiesterase - 5 inhibitors (e.g. Sildenafil, Vardenafil or Tadalafil) and is unable to stop for the duration of the chemoradiotherapy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-01; Primary Completion 2015-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dowell, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Dallas Veterans Affairs Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult men and women otherwise eligible for medical care at Dallas VA Medical center were identified as they presented for consideration of standard therapy.
Groups:
- Nitroglycerin 0.2mg/hr Cohort 1: Nitroglycerin: 0.2mg/hr nitroglycerin transdermal patch daily
- Nitroglycerin 0.4mg/hr Cohort 2: Nitroglycerin: 0.4mg/hr nitroglycerin transdermal patch daily
- Nitroglycerin: 0.6mg/hr Cohort 3: Nitroglycerin: 0.6mg/hr nitroglycerin transdermal patch daily
Period: Overall Study
Arm/Group | Nitroglycerin 0.2mg/hr Cohort 1 | Nitroglycerin 0.4mg/hr Cohort 2 | Nitroglycerin: 0.6mg/hr Cohort 3
Started | 7 | 3 | 3
Completed | 7 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Dose escalation trial of Nitroglycerin: 0.2mg/hr nitroglycerin transdermal patch daily
- Cohort 2: nitroglycerin: 0.4 mg/hr nitroglycerin transdermal patch daily
- Cohort 3: nitroglycerin: 0.6 mg/hr nitroglycerin transdermal patch daily
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 7 | 3 | 3 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 1 | 2 | 8
  >=65 years | 2 | 2 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants] — Population: After extensive effort to locate the raw data so that we can stratify by different cohorts, we were not able to get this data.
  Participants
    Female | 0 | 0 | 0 | 0
    Male | 7 | 3 | 3 | 13
Region of Enrollment [Number; unit: participants]
  United States | 7 | 3 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Experiencing Dose Limiting Toxicities (DLT)
Description: DLT was defined as greater or equal to two instances of grade 3 toxicity, or a single event of grade 4-5 toxicity deemed probably or definitely related to the addition of transdermal neoadjuvant chemoradiation to the standard neoadjuvant chemoradiation
Time Frame: Up to 4-6 weeks for each dosing cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 7 | 3 | 3
Participants | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With a Pathological Complete Response (pCR)
Description: pathological complete response (pCR) at time of surgery following the completion of neoadjuvant therapy. This will be compared to the institutional historical pCR rate.
  Pathologic complete response indicates a complete absence of cancer at the time of surgical resection.
Time Frame: Time of surgery (~ 6-9 wks) following the completion of neoadjuvant therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 7 | 3 | 3
Participants | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: From the first clinic visit to 4-12 weeks after surgery or until resolution of all acute side effects from radiation had occurred, approximately 5 years
Description: investigator assessment, regular laboratory testing
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/7 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=7) | Cohort 2 (N=3) | Cohort 3 (N=3)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=7) | Cohort 2 (N=3) | Cohort 3 (N=3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3)
Grade 3 Headache (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (7) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
GGT Elevation (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hand/Foot Syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Endocrine disorders) | 1 (3) | 0 (0) | 0 (0)
Hypokalmia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Mucositis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Nausea/Vomitting (Gastrointestinal disorders) | 3 (8) | 0 (0) | 0 (0)
Orthostatic Hypotension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity (General disorders) | 3 (3) | 0 (0) | 0 (0)
Radiation Proctitis (General disorders) | 3 (7) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 2 (2) | 0 | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No